CLINICAL TRIAL: NCT00376935
Title: A Double Blind Phase II Study of Multiple Doses of Palifermin (rHuKGF) for the Treatment of Inadequate CD4+ Lymphocyte Recovery in Subjects on Potent Antiretroviral Therapy With Plasma HIV-1 RNA Levels of 200 Copies Per Milliliter or Less
Brief Title: Effectiveness of Palifermin in Increasing CD4 Counts in Treatment-Experienced HIV Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5212; 10147 (Registry Identifier: DAIDS ES); ACTG A5212
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Fibroblast Growth Factor 7

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- 1 (Placebo Comparator): Participants will receive palifermin placebo injection on Days 1, 2, and 3
  Interventions: Drug: Palifermin placebo
- 2 (Experimental): Participants will receive palifermin 20 mcg/kg injection on Days 1, 2, and 3
  Interventions: Drug: Palifermin
- 3 (Experimental): Participants will receive palifermin 40 mcg/kg injection on Days 1, 2, and 3
  Interventions: Drug: Palifermin
- 4 (Experimental): Participants will receive palifermin 60 mcg/kg injection on Days 1, 2, and 3
  Interventions: Drug: Palifermin

INTERVENTIONS:
Drug: Palifermin — Keratinocyte growth factor administered via injection
  Other Names: rHuKGF
  Arms: 2; 3; 4
Drug: Palifermin placebo — Keratinocyte growth factor placebo administered via injection
  Other Names: rHuKGF placebo
  Arms: 1

SUMMARY:
Palifermin is a modified version of a naturally occurring human growth factor that is currently approved by the FDA to treat blood cancers. The purpose of this study is to determine whether palifermin can increase CD4 counts in treatment-experienced HIV infected adults.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) has dramatically improved the clinical outcome for HIV infected adults; however, some people on potent ART experience poor recovery of CD4 counts despite maximum suppression of viral load. Such uncontrolled HIV infection is associated with the reduced ability by the human body to create new T cells (or thymopoiesis). HIV infected adults experiencing reduced thymopoiesis are at increased risk of clinical disease progression.

The thymus is the primary site for CD4 cell development; research suggests that keratinocyte growth factor (KGF) may enhance thymus activity in individuals who exhibit reduced thymopoiesis. Palifermin is a modified version of the naturally occurring KGF that is approved to treat people with hematologic malignancies. The purpose of this study is to evaluate the safety and efficacy of palifermin in increasing CD4 counts, through enhanced thymopoiesis, in treatment-experienced HIV infected adults with suppressed viral loads but low CD4 counts.

This study will last 24 weeks. Participants will be randomly assigned to one of four arms:

* Arm A participants will receive placebo
* Arm B participants will receive palifermin 20 mcg/kg
* Arm C participants will receive palifermin 40 mcg/kg
* Arm D participants will receive palifermin 60 mcg/kg

Participants will receive intravenous doses of their assigned intervention on Days 1, 2, and 3. All participants must remain on their current ART regimen for the duration of the study. ART will not be provided by the study. There will be six study visits, and they will occur at Weeks 1, 2, 4, 8, 12, and 24. All visits will include a targeted physical exam and blood and urine collection.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Receiving potent ART, defined as a combination of three or more antiretroviral drugs for at least 6 months prior to study entry
* CD4 count of 200 cells/mm3 or less within 30 days prior to study entry
* Documented CD4 count obtained at study screening
* Documented current, persistent viral load less than or equal to 200 copies/ml for at least 6 months prior to study entry
* Willing to use acceptable forms of contraception for the duration of the study

Exclusion Criteria:

* Active pancreatitis
* Androgens, Immunomodulators (e.g., growth factors, systemic corticosteroids, HIV vaccines, immune globulin, interleukins, interferons), or investigational ART within 30 days prior to study entry
* Systemic cancer chemotherapy within 30 days prior to study entry, or history of radiation therapy to the neck and chest regions at any time.
* Allergy or sensitivity to any component of palifermin
* Prior treatment with palifermin or other keratinocyte growth factors
* Current drug or alcohol use that, in the opinion of the investigator, may interfere with study participation
* Serious illness or recent surgery that requires systemic treatment or hospitalization. Participants who have completed therapy or are clinically stable on therapy for at least 30 days prior to study entry are not excluded.
* Active cancer
* HIV-1 RNA levels >200 copies/mL within 6 months prior to study entry
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-12; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Jacobson, MD, Study Chair — Division of Infectious Diseases and HIV Medicine, Drexel University College of Medicine
Locations (22):
- United States (22):
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Bmc Actg Crs, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Trillium Health ACTG CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Aiuti F, Mezzaroma I. Failure to reconstitute CD4+ T-cells despite suppression of HIV replication under HAART. AIDS Rev. 2006 Apr-Jun;8(2):88-97. PMID 16848276
- [Background] Franco JM, Rubio A, Martinez-Moya M, Leal M, Merchante E, Sanchez-Quijano A, Lissen E. T-cell repopulation and thymic volume in HIV-1-infected adult patients after highly active antiretroviral therapy. Blood. 2002 May 15;99(10):3702-6. doi: 10.1182/blood.v99.10.3702. PMID 11986226
- [Background] van den Brink MR, Alpdogan O, Boyd RL. Strategies to enhance T-cell reconstitution in immunocompromised patients. Nat Rev Immunol. 2004 Nov;4(11):856-67. doi: 10.1038/nri1484. PMID 15516965
- [Background] Ye P, Kourtis AP, Kirschner DE. Reconstitution of thymic function in HIV-1 patients treated with highly active antiretroviral therapy. Clin Immunol. 2003 Feb;106(2):95-105. doi: 10.1016/s1521-6616(02)00024-4. PMID 12672400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at 22 sites around the States, between February 2007 to April 2008.
Pre-assignment Details: All randomized participants got at least one injection on each of three consecutive days.
Groups:
- Palifermin Placebo: Participants will receive 3 placebo for palifermin IV bolus injections on each of 3 consecutive days: day 1 (entry), day 2 and day 3.
- Palifermin (20 mcg/kg): Participants will receive 1 palifermin 20 mcg/kg (0.004) mL/kg IV bolus injection, two placebo for palifermin IV bolus injections on each of 3 consecutive days: day 1 (entry), day 2 and day 3.
- Palifermin (40 mcg/kg): Participants will receive 1 palifermin 40 mcg/kg (0.008) mL/kg IV bolus injection, two placebo for palifermin IV bolus injections on each of 3 consecutive days: day 1 (entry), day 2 and day 3.
- Palifermin (60 mcg/kg): Participants will receive 1 palifermin 60 mcg/kg (0.012) mL/kg IV bolus injection, two placebo for palifermin IV bolus injections on each of 3 consecutive days: day 1 (entry), day 2 and day 3.
Period: Overall Study
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Started | 25 | 25 | 25 | 24
Completed | 25 | 25 | 25 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg) | Total
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 99
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 (7.8) [42 to 50] | 49 (8.8) [43 to 54] | 45 (9.7) [39 to 54] | 50 (8.9) [46 to 57] | 49 (8.9) [42 to 55]
Age, Customized [Number; unit: participants]
  Between 18 and 29 years | 0 | 0 | 1 | 0 | 1
  Between 30 and 39 years | 4 | 1 | 6 | 2 | 13
  Between 40 and 49 years | 13 | 12 | 8 | 9 | 42
  Between 50 and 59 years | 4 | 8 | 7 | 8 | 27
  Over 60 years | 4 | 4 | 3 | 5 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 1 | 9
  Male | 22 | 23 | 22 | 23 | 90
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 15 | 13 | 12 | 12 | 52
  Black Non-Hispanic | 6 | 9 | 4 | 6 | 25
  Hispanic (Regardless of Race) | 3 | 3 | 8 | 6 | 20
  Asian, Pacific Islander | 1 | 0 | 0 | 0 | 1
  Missing/ Unknown | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 24 | 99
IV drug use [Number; unit: participants]
  Never | 20 | 22 | 19 | 20 | 81
  Previously | 5 | 3 | 6 | 4 | 18
CD4 count [Median (Inter-Quartile Range); unit: cell/mm^3] | 147 [110 to 180] | 155 [126 to 194] | 156 [116 to 197] | 152 [112 to 192] | 153 [116 to 194]
CD8 count [Median (Inter-Quartile Range); unit: cell/mm^3] | 638 [394 to 887] | 615 [464 to 722] | 716 [575 to 999] | 761 [502 to 1099] | 665 [467 to 954]
HIV-1 RNA Categorical [Number; unit: participants]
  < 50 copies/mL | 22 | 22 | 23 | 24 | 91
  = 52 copies/mL | 1 | 0 | 0 | 0 | 1
  = 77 copies/mL | 1 | 0 | 0 | 0 | 1
  = 81 copies/mL | 1 | 0 | 0 | 0 | 1
  = 84 copies/mL | 0 | 0 | 1 | 0 | 1
  = 88 copies/mL | 0 | 1 | 0 | 0 | 1
  = 97 copies/mL | 0 | 1 | 0 | 0 | 1
  = 69440 copies/mL | 0 | 1 | 0 | 0 | 1
  Missing | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Absolute CD4+ Lymphocyte Counts From Baseline (Average of Pre-entry and Entry Values)
Description: Median and inter-quartile range of the change in absolute CD4 count from baseline to study week 12 were calculated for each treatment arm. Baseline CD4+ count was defined as the average of pre-entry and entry CD4 count. If one evaluation was missing, the other one was used. If a subject missed a week 12 CD4 count evaluation, then the CD4 count evaluation obtained after starting study treatment and closest in time to week 12 (using the earlier evaluation if necessary to break a tie) was used in place of the missing week 12 evaluation.
Time Frame: Pre-entry, entry, study week 12
Population: Numbers presented use the intent-to-treat.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Number analyzed (Participants) | 25 | 25 | 25 | 24
cells/mm^3 | 15 [-16 to 23] | 11 [2 to 32] | 12 [-2 to 25] | 8 [-13 to 35]
Statistical Analysis 1: Comparison: Palifermin Placebo vs Palifermin (20 mcg/kg); The null hypothesis is that the distribution of the change in absolute CD4+ lymphocyte counts from baseline to week 12 is the same in the placebo arm and palifermin (20 mcg/kg) arm. The 1-sided alternative hypothesis is that the endpoint distribution is shifted higher in the palifermin (20 mcg/kg) arm; Test type: Superiority or Other; p = 0.1996, Wilcoxon (Mann-Whitney) — P-value reported here was not adjusted for multiple comparisons. A 98.4% confidence upper bound for the shift parameter for each comparison adjusted the multiple comparison issues and restricted the familywise Type I error rate at 0.05; One-sided Wilcoxon rank sum test was used to test the null hypothesis.A 98.4% confidence upper bound for the primary shift parameter was calculated; Shift parameter = -9, 98.4% CI 1-sided [upper limit 14] — The shift parameter (say, X), was calculated as the difference between the distribution of the primary endpoint in the placebo arm and that of in the palifermin arm. X<0 indicates that palifermen is beneficial
Statistical Analysis 2: Comparison: Palifermin Placebo vs Palifermin (40 mcg/kg); The null hypothesis is that the distribution of the change in absolute CD4+ lymphocyte counts from baseline to week 12 is the same in the placebo arm and palifermin (40 mcg/kg) arm. The 1-sided alternative hypothesis is that the endpoint distribution is shifted higher in the palifermin (40 mcg/kg) arm; Test type: Superiority or Other; p = 0.3135, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Shift parameter = -4, 98.4% CI 1-sided [upper limit 17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Palifermin Placebo vs Palifermin (60 mcg/kg); The null hypothesis is that the distribution of the change in absolute CD4+ lymphocyte counts from baseline to week 12 is the same in the placebo arm and palifermin (60 mcg/kg) arm. The 1-sided alternative hypothesis is that the endpoint distribution is shifted higher in the palifermin (60 mcg/kg) arm; Test type: Superiority or Other; p = 0.3662, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Shift parameter = -4, 98.4% CI 1-sided [upper limit 22] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Qualitative Hepatitis C Virus RNA
Time Frame: At study entry
Measure: Number; unit: participants
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Number analyzed (Participants) | 25 | 25 | 25 | 24
participants
  # of participants who had positive HCV results | 4 | 2 | 1 | 5
  # of participants who had negative HCV results | 21 | 22 | 24 | 19
  # of missing | 0 | 1 | 0 | 0

3. Secondary Outcome: Grade 3 or 4 Toxicity for Signs and Symptoms From Randomization to Week 24
Description: Number of subjects had a grade 3 or 4 toxicity for signs and symptoms. The toxicity grade scale has the following meaning: 1=mild, 2=moderate, 3=severe, 4=life-threatening.
Time Frame: From randomization to week 24
Population: Numbers presented use the intent-to-treat approach (i.e. ignoring changes from randomized treatment).
Measure: Number; unit: participants
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Number analyzed (Participants) | 25 | 25 | 25 | 24
participants | 2 | 4 | 2 | 1

4. Secondary Outcome: Change in Naive CD4+ Cell Counts From Randomization
Time Frame: randomization, day 2, study weeks 1, 2, 4, 8, 12 and 24
Population: This analysis was based on observed data only. No imputation was done for missing values. The number of participants with results available varies by study week for each treatment arm.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Number analyzed (Participants) | 25 | 25 | 25 | 24
cells/mm^3
  Day 2 naive CD4+ change: number analyzed (Participants) | 24 | 24 | 22 | 22
  Day 2 naive CD4+ change | -2 [-5 to 2] | -2 [-10 to 3] | -1 [-4 to 2] | -2 [-6 to 1]
  Week 1 naive CD4+ change: number analyzed (Participants) | 24 | 25 | 25 | 24
  Week 1 naive CD4+ change | 0 [-3 to 4] | -2 [-6 to 2] | -1 [-7 to 2] | -1 [-4 to 2]
  Week 2 naive CD4+ change: number analyzed (Participants) | 23 | 22 | 24 | 23
  Week 2 naive CD4+ change | -1 [-8 to 4] | -1 [-5 to 2] | -1 [-4 to 3] | 0 [-7 to 3]
  Week 4 naive CD4+ change: number analyzed (Participants) | 21 | 24 | 19 | 23
  Week 4 naive CD4+ change | 0 [-2 to 4] | -2 [-4 to 1] | 1 [-4 to 3] | 0 [-3 to 5]
  Week 8 naive CD4+ change: number analyzed (Participants) | 24 | 25 | 21 | 23
  Week 8 naive CD4+ change | 3 [-2 to 7] | 0 [-6 to 3] | 1 [-3 to 5] | 2 [-1 to 7]
  Week 12 naive CD4+ change: number analyzed (Participants) | 23 | 23 | 21 | 23
  Week 12 naive CD4+ change | 1 [-6 to 5] | 1 [-7 to 4] | 1 [-3 to 5] | 0 [-6 to 5]
  Week 24 naive CD4+ change: number analyzed (Participants) | 23 | 20 | 22 | 23
  Week 24 naive CD4+ change | 1 [-1 to 10] | -1 [-7 to 4] | 2 [-4 to 8] | 1 [-4 to 7]

5. Secondary Outcome: Change in CT Thymic Index From Randomization
Description: CT thymic index was evaluated at randomization and study week 12, ranging from 0 to 5 whereby 0 means lack of thymic tissue and an organ entirely replaced by fat, 1 means barely recognizable thymic tissue, 2 means minimal soft tissue, 3 means obvious thymic tissue, 4 means moderate thymic tissue, 5 means thymic mass of possible concern for thymoma. Change in CT thymic index from randomization to study week 12 was calculated for participants with both evaluations. The number of participants in each change group was reported by treatment arm.
Time Frame: randomization, study week 12
Population: Participants who had CT thymus evaluations at both randomization and study week 12.
Measure: Number; unit: participants
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Number analyzed (Participants) | 22 | 22 | 22 | 22
participants
  two-sizes-smaller thymus at week 12 | 1 | 0 | 1 | 0
  one-size-smaller thymus at week 12 | 3 | 6 | 3 | 3
  unchanged thymus from randomization to week 12 | 11 | 12 | 13 | 13
  one-size-larger thymus at week 12 | 7 | 4 | 4 | 6
  two-sizes-larger thymus at week 12 | 0 | 0 | 1 | 0

6. Secondary Outcome: Change in Absolute CD4+ Lymphocyte Counts From Randomization to Day 2, Weeks 1, 2, 4, 8, 12, 24.
Time Frame: randomization, day 2, study weeks 1, 2, 4, 8, 12 and 24
Population: This analysis was based on observed data only. No imputation was done for missing values. NOTE: The number of participants may vary in each study week for each treatment arm. The maximum number for each arm are showed above.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Number analyzed (Participants) | 25 | 25 | 25 | 24
cells/mm^3
  Day 2 CD4+ change | -4 [-15 to 22] | 2 [-13 to 15] | -12 [-28 to 1] | -5 [-21 to 16]
  Week 1 CD4+ change | 1 [-10 to 7] | -12 [-31 to 15] | -9 [-33 to 12] | 6 [-27 to 22]
  Week 2 CD4+ change: number analyzed (Participants) | 24 | 24 | 24 | 24
  Week 2 CD4+ change | -1 [-10 to 37] | 1 [-29 to 9] | 14 [-3 to 21] | 2 [-20 to 26]
  Week 4 CD4+ change: number analyzed (Participants) | 23 | 24 | 23 | 23
  Week 4 CD4+ change | 6 [-17 to 25] | 1 [-17 to 9] | 16 [-15 to 29] | 2 [-35 to 28]
  Week 8 CD4+ change: number analyzed (Participants) | 25 | 25 | 24 | 24
  Week 8 CD4+ change | 10 [-14 to 26] | 2 [-15 to 20] | 20 [-5 to 39] | 9 [-8 to 32]
  Week 12 CD4+ change: number analyzed (Participants) | 24 | 23 | 23 | 24
  Week 12 CD4+ change | 14 [-17 to 27] | 11 [1 to 32] | 12 [-6 to 38] | 8 [-13 to 35]
  Week 24 CD4+ change: number analyzed (Participants) | 25 | 23 | 25 | 24
  Week 24 CD4+ change | 14 [-10 to 26] | 8 [-13 to 34] | 14 [1 to 50] | 15 [0 to 46]

7. Secondary Outcome: Grade 3 or 4 Lab Toxicities From Randomization to Week 24
Description: Number of subjects had a grade 3 or 4 toxicity for laboratory abnormalities. The toxicity grade scale has the following meaning: 1=mild, 2=moderate, 3=severe, 4=life-threatening.
Time Frame: From randomization to study week 24
Measure: Number; unit: participants
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Number analyzed (Participants) | 25 | 25 | 25 | 24
participants | 4 | 5 | 4 | 6

8. Secondary Outcome: Number of Death From Randomization to Week 24
Description: Number of subjects died.
Time Frame: From randomization to week 24
Measure: Number; unit: participants
Arm/Group | Palifermin Placebo | Palifermin (20 mcg/kg) | Palifermin (40 mcg/kg) | Palifermin (60 mcg/kg)
Number analyzed (Participants) | 25 | 25 | 25 | 24
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Palifermin Placebo | Palifermin (20 Mcg/kg) | Palifermin (40 Mcg/kg) | Palifermin (60 Mcg/kg)
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25 | 1/25 | 0/24
Other Adverse Events (participants affected / at risk) | 25/25 | 24/25 | 25/25 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin Placebo (N=25) | Palifermin (20 Mcg/kg) (N=25) | Palifermin (40 Mcg/kg) (N=25) | Palifermin (60 Mcg/kg) (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palifermin Placebo (N=25) | Palifermin (20 Mcg/kg) (N=25) | Palifermin (40 Mcg/kg) (N=25) | Palifermin (60 Mcg/kg) (N=24)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 2 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 3 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 2
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 3 | 3
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 3 | 2
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 5 | 0 | 1
Chest pain (General disorders) | 1 | 3 | 0 | 0
Chills (General disorders) | 0 | 3 | 0 | 0
Fatigue (General disorders) | 3 | 5 | 2 | 3
Oedema peripheral (General disorders) | 1 | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 4 | 4 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 7 | 8 | 3 | 5
Blood albumin (Investigations) | 1 | 2 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 3 | 4 | 3
Blood bicarbonate (Investigations) | 4 | 4 | 2 | 2
Blood bilirubin increased (Investigations) | 10 | 6 | 6 | 7
Blood calcium decreased (Investigations) | 4 | 4 | 0 | 2
Blood cholesterol abnormal (Investigations) | 2 | 2 | 0 | 2
Blood creatinine increased (Investigations) | 6 | 1 | 4 | 4
Blood glucose abnormal (Investigations) | 3 | 3 | 3 | 4
Blood glucose decreased (Investigations) | 3 | 5 | 3 | 7
Blood glucose increased (Investigations) | 9 | 13 | 16 | 16
Blood phosphorus decreased (Investigations) | 2 | 3 | 1 | 1
Blood potassium decreased (Investigations) | 2 | 5 | 4 | 4
Blood potassium increased (Investigations) | 1 | 1 | 2 | 0
Blood sodium decreased (Investigations) | 5 | 7 | 7 | 5
Blood sodium increased (Investigations) | 1 | 3 | 1 | 0
Carbon dioxide (Investigations) | 0 | 1 | 2 | 3
Carbon dioxide abnormal (Investigations) | 2 | 4 | 2 | 2
Lipase increased (Investigations) | 1 | 2 | 3 | 2
Neutrophil count decreased (Investigations) | 4 | 2 | 4 | 1
Platelet count decreased (Investigations) | 5 | 5 | 5 | 1
White blood cell count decreased (Investigations) | 3 | 1 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 5 | 6 | 3
Headache (Nervous system disorders) | 1 | 4 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 3 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description:In accordance with the Clinical Trial Agreement between NIAID (DAIDS)and company collaborators,NIAID provides companies with a copy of any abstract,press release,or manuscript prior to submission for publication with sufficient time for company review and comment.The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and 5 business days for abstracts,to preserve U.S. or foreign patent or other intellectual property rights.